CLINICAL TRIAL: NCT02277405
Title: A Comparison of Endotracheal Intubation Using the Shikani Optical Stylet or the Endoeye Flexible Intubation During Pediatric Resuscitation
Brief Title: Pediatric Intubation During Resuscitation
Acronym: PIDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ETI/2014/04
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Intubation; Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation without chest compressions.
  Interventions: Device: Shikani Optical Stylet; Device: Endoeye Flexible Intubation (LF-V)
- Intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of pediatric mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: Shikani Optical Stylet; Device: Endoeye Flexible Intubation (LF-V)

INTERVENTIONS:
Device: Shikani Optical Stylet — Optical intubation
Device: Endoeye Flexible Intubation (LF-V) — endoscopy intubation

SUMMARY:
The aim of the study was to compare time and success rates of four intubation devices in a cardiopulmonary scenario with and without chest compressions with a standardized pediatric manikin model.

DETAILED DESCRIPTION:
Emergency airway management during resuscitation is a critical skill in emergency medicine. According to the European Resuscitation Council (ERC) guidelines for resuscitation 2010 , endotracheal intubation (ETI) is considered the gold standard during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (paramedics, nurses, physicians)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | 1 month
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 month
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
VAS score | 1 month
  participants were asked which method they would prefer in a real-life resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland